CLINICAL TRIAL: NCT06529848
Title: Ischemia With No Obstruction of Coronary Arteries: Underlying Mechanisms and the Impact of Exercise Training (EXINOCA)
Brief Title: Impact of Exercise Training on Ischemia With Non-Obstructive Coronary Arteries (INOCA): The ExINOCA Study
Acronym: ExINOCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Eva Prescott, MD Clinical Professor, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ExINOCA
Record Dates: First submitted 2024-07-04; First posted 2024-07-31 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Coronary Microvascular Disease; CMD
MeSH Terms: conditions — Microvascular Angina | interventions — Exercise; Endurance Training

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial in which 100 angina patients with reduced flow reserve (INOCA patients) are randomized 1:1 to either exercise training or control (no exer-cise training).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Active Comparator): The exercise intervention consists of supervised training 40-50 minutes x 3 weekly for 12 weeks.
  Interventions: Other: Exercise training
- Control (No Intervention): The participants who are randomized to the no-training group will be offered exercise train-ing after the intervention is completed. Participants will be encouraged to not change their lifestyle or medication throughout the study period.

INTERVENTIONS:
Other: Exercise training — The training sessions are consist of cycling and as follows: a 10 min warm-up at a light intensity, 20-35 min of cycling exercise in intervals at varying intensities from light (~60% of max heart rate) to more intensive (80-90% of max heart rate) and ending with 5 min of warm-down at a light intensity. The training intensity will be progressive during the course of the intervention period. The cycling training sessions are supervised .
  Home training is allowed up to once a week if participants are able to adhere to the prescribed intensity levels.
  Training sessions are closely monitored to ensure effectiveness and safety. This includes heart rate monitoring, perceived exertion assessment.
  Other Names: Physical activity; Endurance training
  Arms: Exercise

SUMMARY:
The purpose of the study is to identify causes of chest pain in patients experiencing chest pain with no signs of narrowing of the coronary arteries of the heart, and to investigate whether physical exercise can improve coronary microvascular function.

Hypotheses:

The first hypothesis is that in INOCA, with reduced function of microvasculature of the heart, this reduced function also occurs in other organs of the body.

The second hypothesis is that regular physical activity (aerobic exercise training) can improve coronary microvascular function, reduce symptoms, and that there is a parallel improvement in vascular function in other organs of the body.

DETAILED DESCRIPTION:
A significant number of patients suspected of chronic coronary syndrome do not have coronary artery obstruction and in a large proportion of these, their symptoms are attributed to coronary microvascular dysfunction (CMD), a condition known as ischemia with no obstructive coronary artery disease (INOCA). Despite a considerable patient population affected by INOCA, the specific mechanisms underlying CMD are not fully understood, often resulting in a lack of targeted treatment. There is evidence to suggest that exercise capacity is linked to coronary microvascular function, positing that exercise training could potentially reverse microvascular dysfunction and address its mechanistic origins, a hypothesis yet to be explored.

This study aims to identify mechanisms underlying CMD in angina and to assess whether exercise training can improve the condition.

The current study is a randomized controlled trial testing the effect of exercise training in patients with CMD. 100 patients will be randomized 1:1 to exercise training or control. The primary outcome is coronary microvascular function, secondary outcomes include symptoms and microvascular function in cutaneous tissue, skeletal muscle, and adipose tissue.

ELIGIBILITY:
Inclusion Criteria:

* Coronary microvascular dysfunction, defined as myocardial bloodflow reserve (MBFR) < 2.5 or hyperemic myocar-dial blood flow (hMBF)<2.3 ml/g/min using [15O]H2O-PET
* No obstructive coronary artery disease

Exclusion Criteria:

* Females of childbearing potential (defined as a premeno-pausal female capable of becoming pregnant). The female patient must either be postmenopausal, defined as amen-orrhea for at least 1 year, or surgically sterile
* Heart failure, defined as left ventricular ejection fraction of less than 40%
* Uncontrolled hypertension defined as blood pressure above target 140/90 for all
* Co-morbidity resulting in <1 year expected survival
* Considered by the investigator, for any reason, to be an un-suitable candidate for the study.
* Unable or unwilling to exercise, e.g. due to arthritis or in-jury*
* Already are regularly physically active and/or have a maxi-mal oxygen uptake >45 ml/kg/min

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
Change in Myocardial Blood Flow Reserve (MBFR) | From baseline and after 3 months
  Change in MBFR assessed by [15O]H2O-PET-scan

SECONDARY OUTCOMES:
Change in symptom burden assessed by Seattle Angina Questionnaire | From baseline and after 3 months
  Seattle angina questionnaire/selfreported (scale range 0-100, 0=poor and 100=excellent health status)
Change in exercise capacity | From baseline and after 3 months
  Oxygen uptake during exhaustive exercise
Change in global rest perfusion in patients with angina symptoms and CMD | From baseline and after 3 months
  Change in Myocardial Blood Flow assessed by [15O]H2O-PET-scan
Change in global stress perfusion in patients with angina symptoms and CMD | From baseline and after 3 months
  Change in hyperemic Myocardial Blood Flow assessed by [15O]H2O-PET-scan

OTHER OUTCOMES:
Vascular Function Adaptations | From baseline and after 3 months
  Changes in Arterial compliance (C = ΔV/ ΔP) calculated from intraarterial pressure ΔP and arterial diameter (ΔD) measured by ultrasound Doppler
Changes in skin microvascular function | From baseline and after 3 months
  Hand microcirculatory blood flow assessed by Laser Speckle Contrast Imaging
Change in plasma levels of markers related to vascular function | From baseline and after 3 months
  Plasma levels of markers related to vascular function assessed by Mesoscale/ELISA
Changes in Arterial Blood Pressure | From baseline and after 3 months
  Assessed by automated blood pressure at rest
Change in plasma Lipids | From baseline and after 3 months
  Conducted through clinical chemical analysis to measure levels of HDL, and triglycerides in the blood, providing insights into lipid profiles.
Changes in Plasma Levels of Inflammatory Markers | From baseline and after 3 months
  Measured using Mesoscale/ELISA/O-Link platforms to evaluate the presence and levels of inflammatory markers, indicating systemic inflammation.
Proteomic and transcriptomic analyses | From baseline and after 3 months
  Changes in gene and protein expressions patterns in small arteries

CONTACTS AND LOCATIONS:
Overall Officials: Eva Prescott, MD, DMSc, Principal Investigator — University of Copenhagen; Ylva Hellsten, Principal Investigator — University of Copenhagen
Locations (2):
- Denmark (2):
  - Frederiksberg Hospital, Dept. of Cardiology, Building 16, Y3, Nordre Fasanvej 57, Frederiksberg, Denmark, 2000, Copenhagen
  - Frederiksberg Hospital, Dept. of Cardiology, Building 16, Y3, Nordre Fasanvej 57, Frederiksberg

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-29): https://cdn.clinicaltrials.gov/large-docs/48/NCT06529848/Prot_SAP_000.pdf